CLINICAL TRIAL: NCT01828398
Title: tDCS and Robotic Therapy in Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, MD, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Stroke_tDCS
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Stroke; Upper Extremity Impairments
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sham-tDCS + UE robot-assisted therapy (Sham Comparator): This group will receive the same robot-assisted therapy of the intervention group, in association of sham-tDCS. This consists in a 30 seconds stimulation, with the same instrumentation and electrodes placement. This method of sham stimulation was previously validated.
  Interventions: Device: sham-tDCS + UE robot-assisted therapy
- real-tDCS + UE robot-assisted therapy (Experimental): This group will receive continuous stimulation lasting 30 minutes during the session of robot-assisted therapy. The training session, which includes multiplanar, repetitive and target reaching movements, will be given 5 times a week for 2 weeks(REO Therapy System; Motorika, Medical LTD, Israel). Each session will last about 30 minutes.
  Transcranial direct current stimulation (tDCS) will be administered as follows. The anode will be placed on the primary motor cortex (M1) of the affected hemisphere and the cathode on the contralateral M1 area. The direct current is transmitted through a pair of sponge electrodes, with a surface of 35 cm2 (7x5), soaked in saline solution and, it is generated by a constant current stimulator, with rechargeable batteries (Brainstim, EMS, Italy). This continuous stimulation lasted 30 minutes, with an intensity of 1mA.
  Interventions: Device: real-tDCS + UE robot-assisted therapy

INTERVENTIONS:
Device: real-tDCS + UE robot-assisted therapy
  Arms: real-tDCS + UE robot-assisted therapy
Device: sham-tDCS + UE robot-assisted therapy
  Arms: sham-tDCS + UE robot-assisted therapy

SUMMARY:
After stroke a limited motor recovery in the paretic upper limb accounts for a large proportion of the disabling sequelae. Only about 15% of those with initial complete upper limb paralysis after stroke recover functional use of their impaired arm in daily life.

The aim of this study is to test the effects of tDCS combined with upper extremity robot-assisted therapy on stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Males and females subjects. Age > 18 years.
* Diagnosis of first ischemic stroke
* Impairment of the upper limb
* Trunk control defined in the Trunk-Control Test (TCT), with a score > 50.

Exclusion Criteria:

* anyone who does not have adequate understanding of verbal or written information in Italian sufficient to complete any test
* Impaired cognitive functioning: score less than 24 on the Mini Mental Status Examination (MMSE)
* contraindications to single-pulse transcranial magnetic stimulation (TMS)(TMS will be used to measure cortical excitability): presence of a history of epilepsy, frequent headaches or neck pain, implantable devices (ventriculoperitoneal shunts, pacemakers, intrathecal pumps, intracranial metal implants)
* Contraindications to tDCS: intracranial metal implants that can be stimulated, incorrectly positioned or over-heated by the electric current
* Neurological or psychiatric pathology
* severe cardio-pulmonary, renal, hepatic diseases
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity | A week prior to treatment beginning
  Measure of upper extremity motor impairment. The upper extremity score ranges from 0-66.

SECONDARY OUTCOMES:
Box and Block Test | A week prior to treatment beginning
  Test for gross motor function. It counts the number of blocks that can be transported from one compartment of a box to another compartment within 1 minute.
Ashworth Modified Scale | A week prior to treatment beginning
  a 6 point measure of spasticity. We will assess the spasticity at the shoulder, elbow and, wrist
Motor Activity Log (MAL) | A week prior to treatment beginning
  Assessment of the change in real-world arm use in activities of daily living. Subjects are asked to score the quality of movement as well as amount of use of the affected arm in a number of common daily activities.
Assessment of cortical excitability (TMS) | A week prior to treatment beginning
  MEP of upper limb muscles (first dorsal interosseous) will be recorded with surface EMG electrodes. neurophysiological parameters analyzed:
  * motor threshold at rest
  * MEP recruitment curve at rest
  * MEP amplitude

CONTACTS AND LOCATIONS:
Locations (1):
- Ferrara University Hospital, Ferrara, Italy

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411